CLINICAL TRIAL: NCT01279252
Title: A Phase II Trial of Broad Spectrum Antibiotic Therapy for Early Stage, Non-progressive Chronic Lymphocytic Leukaemia Without Adverse Prognostic Factors
Brief Title: CLL Empirical Antibiotic Regimen
Acronym: CLEAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Dr Stephen Devereux, King's College Hospital NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLEAR
Record Dates: First submitted 2011-01-17; First posted 2011-01-19 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2015-09

CONDITIONS: Chronic Lymphocytic Leukaemia (CLL)
MeSH Terms: conditions — Leukemia, B-Cell | interventions — Metronidazole; Clarithromycin; Ciprofloxacin; Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antibiotic regimen (Experimental)
  Interventions: Drug: metronidazole, clarithromycin, ciprofloxacin and lansoprazole

INTERVENTIONS:
Drug: metronidazole, clarithromycin, ciprofloxacin and lansoprazole

SUMMARY:
The purpose of this study is to evaluate whether patients with previously untreated, early stage CLL respond to empirical broad spectrum antibiotics and therefore test the hypothesis that occult bacterial infections are involved in the induction and maintenance of CLL.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* ECOG performance status of 2 or less.
* CLL with a diagnostic score of 4 or 5.
* Clinical stage A disease.
* No disease progression over a minimum of 1 month prior to commencement of therapy.
* Less than 2 adverse prognostic factors.
* Absence of adverse cytogenetics.
* Expected survival > 6 months.
* Able to give informed consent.
* No clinical evidence of active infection at the time of study entry.
* No known allergy to any of the study medications.
* Renal and liver function tests within normal limits.

Exclusion Criteria:

* Disease progression during screening period.
* Known positivity for HIV types 1 or 2.
* Active infection at the time of screening.
* Pregnancy or lactation.
* Females of childbearing potential† and males not willing to practice an effective method of contraception whilst receiving the antibiotic regimen and for 4 weeks after the last dose.
* Concomitant medication likely to produce serious interaction with study drugs including warfarin type oral anticoagulants and anti-epileptics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2011-07; Primary Completion 2015-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Overall response rate [Complete Remission (CR) + Partial Remission (PR)] | 6 months

SECONDARY OUTCOMES:
Incidence of CTCAE grade 2 or above treatment related toxicity | From day 1 to 6 weeks
Bone marrow Minimal Residual Disease (MRD) status in patients who achieve CR | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Devereux, PhD, FRCP, FRCPath, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom